CLINICAL TRIAL: NCT01093755
Title: Does Intensive Acid Suppression Reduce Esophageal Inflammation and Recurrent Barrett's Esophagus Following Ablation?: A Randomized Controlled Trial
Brief Title: Does Intensive Acid Suppression Reduce Esophageal Inflammation and Recurrent Barrett's Esophagus Following Ablation?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Prasad G. Iyer, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-007252
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Inflammation; Barrett's Esophagus
Keywords: Barrett's Esophagus; Radiofrequency ablation; Patients post-radiofrequency ablation for Barrett's Esophagus.
MeSH Terms: conditions — Inflammation; Barrett Esophagus | interventions — Dexlansoprazole; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexlansoprazole (Active Comparator): Participants will be treated with dexlansoprazole 60-90 mg/day for 6 months
  Interventions: Drug: dexlansoprazole
- omeprazole (Active Comparator): Participants will be treated with omeprazole 20mg/day for a minimum of 6 weeks. If symptomatic can increase dose by 20mg twice.
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: dexlansoprazole — Intensive acid suppression with dexlansoprazole 60-90 mg/day for 6 months
  Other Names: Dexilant
  Arms: dexlansoprazole
Drug: Omeprazole — Escalating doses of omeprazole (20-60 mg/day) for 6 months
  Other Names: Prilosec
  Arms: omeprazole

SUMMARY:
The investigators hypothesize that intensive acid suppression with a long acting high potency proton pump inhibitor (PPI) drug dexlansoprazole will lead to a greater decrease in levels of inflammatory mediators (compared to conventional PPIs) in the esophagus, which could potentially lead to decreased recurrence of intestinal metaplasia following endoscopic ablation.

DETAILED DESCRIPTION:
Patients who achieve complete remission of intestinal metaplasia following ablation will be randomized (using concealed allocation, like the flip of a coin) to either intensive acid suppression with dexlansoprazole 60-90 mg/day or to symptom guided acid suppression with escalating doses of omeprazole (20-60 mg/day) for 6 months. Control of reflux will be assessed using 24 hour ambulatory pH monitoring. The need to escalate drug dosage at the 3 month visit will be determined by presence of excessive acid exposure on ambulatory pH monitoring. Biopsies of esophageal tissue will be obtained at baseline, then at 3 months and 6 months following randomization to measure changes in inflammatory biomarkers.

ELIGIBILITY:
Patients who have undergone ablation for Barrett's Esophagus (BE) and High Grade Dysplasia (HGD) or Low Grade Dysplasia (LGD) with Photodynamic Therapy (PDT)/Radiofrequency ablation and endoscopic mucosal resection who have no endoscopic and histologic evidence of specialized intestinal metaplasia on biopsies from the esophagus on two successive endoscopies post ablation will be offered enrollment in the study.

Inclusion criteria:

1. Absence of intestinal metaplasia on endoscopy (under Narrow Band Imaging) and on histology (from biopsies taken from gastroesophageal junction and distal esophagus) on two successive surveillance endoscopies.
2. Able to consent to study
3. Males and females age 18-90
4. Life expectancy of 5 years or greater.

Exclusion criteria:

1. Pregnancy
2. Inability to consent for the procedure
3. Anticoagulation therapy precluding performance of ambulatory pH monitoring and/or biopsies
4. Intolerance to proton pump inhibitors
5. Elevation in Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), (liver enzymes), bilirubin or alkaline phosphatase more than five times the upper limit of normal.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prasad Iyer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Mayo Clinic patients in Rochester, Minnesota who had undergone an ablation procedure for Barrett's Esophagus.
Period: Overall Study
Arm/Group | Dexlansoprazole | Omeprazole
Started | 16 | 14
Completed | 13 | 10
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexlansoprazole | Omeprazole | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (6.9) | 59.1 (8.9) | 61.5 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 14 | 12 | 26
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30
High Grade Dysplasia/Intramucosal Carcinoma [Number; unit: participants]
  Subjects with High-Grade Dysplasia/Carcinoma | 12 | 10 | 22
  Subjects with Low-Grade Dysplasia | 4 | 4 | 8
Body Mass Index [Mean (Standard Deviation); unit: kg/height in meters^2] | 30.9 (3.4) | 29.3 (4.2) | 30.14 (3.84)
Barrett's Esophagus segment length, pre-ablation [Mean (Standard Deviation); unit: cm] | 5.3 (3.5) | 4.8 (4.3) | 5.06 (3.84)
Diaphragmatic Hernia present [Number; unit: Participants]
  Subjects with Diaphragmatic Hernia | 15 | 13 | 28
  Subjects without Diaphragmatic Hernia | 1 | 1 | 2
Diaphragmatic Hernia length [Mean (Standard Deviation); unit: cm] | 3.6 (2.3) | 3.0 (1.7) | 3.3 (2.05)
Number undergoing Endoscopic Mucosal Resection [Number; unit: Participants]
  Subjects undergoing resection | 16 | 12 | 28
  Subjects not undergoing resection | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Inflammation Biomarker Tissue PGE2 Level
Description: Change from baseline in esophageal tissue biopsy prostaglandin E2 (PGE2) level, as determined by enzyme immunoassay
Time Frame: 3 months, 6 months
Measure: Mean (Standard Deviation); unit: nanograms/gram of tissue
Arm/Group | Dexlansoprazole | Omeprazole
Number analyzed (Participants) | 16 | 14
nanograms/gram of tissue
  Change from baseline at 3 months | 1.35 (3.16) | -0.02 (1.47)
  Change from baseline at 6 months | 1.19 (3.58) | -0.06 (1.45)
Statistical Analysis 1: Comparison: Dexlansoprazole vs Omeprazole; Comparison between the two treatment groups at 3 months; Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dexlansoprazole vs Omeprazole; Comparison between the two treatment groups at 6 months; Test type: Superiority or Other; p = 0.52, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Esophageal Inflammation Biomarker COX-2 Gene Expression
Description: Change from baseline in esophageal issue biopsy cyclooxygenase-2 (COX-2) gene expression, as determined by Western blot.
Time Frame: 3 months, 6 months
Measure: Mean (Standard Deviation); unit: % of tubulin
Arm/Group | Dexlansoprazole | Omeprazole
Number analyzed (Participants) | 16 | 14
% of tubulin
  Change from baseline at 3 months | 36.81 (73.55) | 27.17 (176.82)
  Change from baseline at 6 months | 56.54 (98.77) | 25.49 (210.67)
Statistical Analysis 1: Comparison: Dexlansoprazole vs Omeprazole; Comparison between the two treatment groups at 3 months; Test type: Superiority or Other; p = 0.70, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dexlansoprazole; Comparison between the two treatment groups at 6 months; Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Arm/Group | Dexlansoprazole | Omeprazole
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No